CLINICAL TRIAL: NCT00841477
Title: An Hepatitis B Vaccine Model for HIV Vaccine Trials in Drug Users
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Professor of Epidemiology, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: DESPR DA017505
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis B Infection; Hepatitis C Infection; HIV Infection
Keywords: druguser,HB vaccine adherence, HBV, HCV, HIV incidence
MeSH Terms: conditions — Hepatitis B; Hepatitis C; HIV Infections | interventions — Hepatitis B Vaccines; Appointments and Schedules

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A1 (No Intervention): standard behavioral intervention, standard HB vaccine schedule (0,1,6month)
- A2 (Active Comparator): standard behavioral intervention, accelerated HB vaccine schedule (0,1,2month)
  Interventions: Biological: hepatitis B vaccine 3 dose schedule (0,1,2 month)
- B1 (Active Comparator): enhanced behavioral intervention, standard vaccine schedule
  Interventions: Behavioral: HBV Vaccination Self-Efficacy Intervention
- B2 (Active Comparator): enhanced behavioral intervention, accelerated vaccine schedule (0,1,2MONTH)
  Interventions: Biological: hepatitis B vaccine 3 dose schedule (0,1,2 month); Behavioral: HBV Vaccination Self-Efficacy Intervention

INTERVENTIONS:
Biological: hepatitis B vaccine 3 dose schedule (0,1,2 month) — hepatitis B (HB) vaccine: Engerix-B (GlaxoSmithKline) (20 µg/dose) accelerated HB vaccine schedule (0,1,2 month),vs, standard HB vaccine schedule (0,1,6 m)
  Other Names: accelerated HB vaccine schedule
  Arms: A2; B2
Behavioral: HBV Vaccination Self-Efficacy Intervention — HB Vaccination Intervention consists of 4 sessions - Sessions 1, 2: at screening and enrollment after intake, vs regular risk reduction education Sessions 3, 4: coincide with the vaccination schedule ions 4 before 3rd dose
  Other Names: enhanced behavioral intervention
  Arms: B1; B2

SUMMARY:
The goal of the proposed study is to use the HBV vaccine as a model for a future HIV vaccine trial, examining the efficacy of community-based outreach intervention as well as an accelerated vaccine schedule as a method for increasing acceptance/adherence with HBV vaccination protocols among not-in-treatment drug users. This study will also examine the effect of HBV vaccination coupled with community-based outreach intervention on reducing the incidence of HIV, HBV and HCV infections and the frequency of needle use and sexual risk behaviors related to these viral transmissions. A secondary purpose will be to assess the antibody response after HBV vaccination as a measurement of immunological response in drug users.

DETAILED DESCRIPTION:
This project will evaluate an HBV vaccination program as a model for future HIV vaccine efficacy trials in a community-based study of drug users. Two components will be analyzed in an effort to increase vaccine acceptance/adherence - behavioral intervention & an accelerated vaccine schedule. The study also will examine the effect of these variables on risk behaviors and incidence of HIV, HBV, & HCV infections. To accomplish these objectives, we propose a randomized behavioral intervention field trial. We will enroll 1600 current cocaine or heroin users negative for HBV & HIV markers from two closely matched, low-income, high drug endemic communities in Houston. All participants will be offered HBV vaccination and follow-up viral testing. One community will be randomly assigned to receive an outreach behavioral intervention designed to increase vaccine awareness and vaccine compliance. The other community will receive standard care. Participants electing to be vaccinated will be randomized to either a 0,1,6 month or a 0,1,2, month vaccine schedule. Groups will be followed for two years to determine rates of HBV vaccine acceptance/adherence to the 3-dose protocol. We also will measure any changes in risk behaviors & incidence of HIV/HBV/HCV infections as well as HBV vaccine immune response, if vaccinated. Drug users are the largest group of newly diagnosed HIV cases and so creating a model for an HIV vaccine's acceptance and adherence in this population is an important public health goal. This study will serve as a model for future HIV vaccine trials and will provide information on the effectiveness of outreach programs for increasing immunization among drug users. Unless an effective model based upon empirical experience is developed, any attempt to implement a HIV vaccination program among drug users is likely to be frustrated. If HBV vaccination coupled with outreach intervention can reduce risk behaviors and decrease the incidence of HIV/HCV infection, then this study will have a tremendous impact on the current HBV/HIV/HCV prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

* using cocaine/heroin in last 7 days, age over 18 years old from two matched in population size, income and demographic communities, known with high rate of drug using and STD; competent to consent for urine drug screening and viral markers (anti-HIV, HBsAg/anti-HBs, anti-HCV) testing; those negative for HIV/HBV will be contacted for HB vaccination study.

Exclusion Criteria:

* age under 18 or not from the target communities, negative for urine drug test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Actual)
Dates: Start 2004-01; Primary Completion 2007-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
compliance (adherence) for 3 doses hepatitis vaccination | Jan, 2004 - June 2008

SECONDARY OUTCOMES:
incidence of HIV and HCV infection and change of risk behaviors | Jan, 2004- June 2009
immunological response | Feb 2004 - June 2008

CONTACTS AND LOCATIONS:
Overall Officials: Lu-Yu Hwang, MD, Principal Investigator — University of Texas-HSC at Houston
Locations (1):
- University of Texas-HSC at Houston, School of Public Health, Houston, Texas, United States

REFERENCES:
- [Result] Hwang LY, Grimes CZ, Tran TQ, Clark A, Xia R, Lai D, Troisi C, Williams M. Accelerated hepatitis B vaccination schedule among drug users: a randomized controlled trial. J Infect Dis. 2010 Nov 15;202(10):1500-9. doi: 10.1086/656776. Epub 2010 Oct 11. PMID 20936979
- [Result] Tran TQ, Grimes CZ, Lai D, Troisi CL, Hwang LY. Effect of age and frequency of injections on immune response to hepatitis B vaccination in drug users. Vaccine. 2012 Jan 5;30(2):342-9. doi: 10.1016/j.vaccine.2011.10.084. Epub 2011 Nov 8. PMID 22075088
- [Result] Shah DP, Grimes CZ, Brown E, Hwang LY. Demographics, socio-behavioral factors, and drug use patterns: what matters in spontaneous HCV clearance? J Med Virol. 2012 Feb;84(2):235-41. doi: 10.1002/jmv.22271. PMID 22170543
- [Result] Grimes CZ, Hwang LY, Wei P, Shah DP, Volcik KA, Brown EL. Differentially regulated gene expression associated with hepatitis C virus clearance. J Gen Virol. 2013 Mar;94(Pt 3):534-542. doi: 10.1099/vir.0.047738-0. Epub 2012 Nov 14. PMID 23152368
- [Result] Kamath GR, Shah DP, Hwang LY. Immune response to hepatitis B vaccination in drug using populations: a systematic review and meta-regression analysis. Vaccine. 2014 Apr 25;32(20):2265-74. doi: 10.1016/j.vaccine.2014.02.072. Epub 2014 Mar 12. PMID 24631093
- [Result] Lu-Yu. Hwang*, Carolyn. Grimes "Human Immunodeficiency Virus, hepatitis B and C Virus infections among injecting and non-injecting drug users from inner city neighborhoods " Insight and Control of Infectious Disease in Global Scenario, Priti Kumar Roy (Ed), ISBN 978-953-51-0319-6, 2012, p45-60 InTech, Available from http://www.intechopen.com/articles/show/title/immunodeficiency-virus-hepatitis-b-and-hepatitis-c-virus-infections-among-injecting-and-non-injectin